CLINICAL TRIAL: NCT05348798
Title: Assessment of Personality Traits Associated With Exercise Addiction in Ultra Endurance Athletes
Brief Title: Personality Traits and Exercise Addiction in Ultra Endurance Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: INSERM UMR U1075 Comète GIP Cyceron, unicaen, Caen Normandie (Unknown)
Responsible Party: Principal Investigator, Joffrey DRIGNY, MD MSc, Attending physician in Sport Medicine and PM&R departments, University Hospital, Caen
Other Study IDs: UltrAddict 3363
Record Dates: First submitted 2022-04-16; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Exercise Addiction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultra endurance athletes: Individual participating in ultra endurance sports (events exceeding 6 hours) including running, cycling, triathlon, swimming and Nordic skiing. Participants are above 18 years of age and volunteer to participate in this web-based survey.
  Interventions: Other: Web based survey

INTERVENTIONS:
Other: Web based survey — Web-based survey on exercise addiction and personality traits

SUMMARY:
Ultra endurance sports (events exceeding 6 hours) is becoming increasingly popular and Exercise Addiction (EA) is frequent in this type of sports, which are characterized by very high training volume. However, little is known about the personality traits of athletes who are more likely to develop EA. This study aims to assess the personality traits associated with EA in ultra endurance athletes. We designed a cross sectional study. Participants have to fill a web-based questionnaire including the Big Five Personality Test for assessing the personality traits and the Exercise Dependence Scale-Revised (EDS-R) for assessing EA. Also they have to fill a personal question about demographics (age, gender, work), sport practice and eating habits. A minimum sample size of 300 participants is expected. Statistical analyses will test the association between personality traits and the presence (or absence) of EA according to the EDS-R. Secondary analysis will test the association between the type of sport (running, cycling, triathlon, swimming), the volume of sport practice and the presence of eating disorders and EA.

ELIGIBILITY:
Inclusion Criteria:

* athletes participating in ultra endurance sport events (exceeding 6 hours) in running/trail, cycling, swimming, Nordic skiing
* individuals who volunteered to participate in the study
* individuals with access to internet
* Individuals reading French

Exclusion Criteria:

* individuals not meeting the inclusion criterias
* individuals who did not participate in an ultra endurance event in the previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All ultra endurance athletes who volunteered to participate in the survey
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Exercise Addiction | One single evaluation at a single point in time through study completion, an average of 3 months
  The Exercise Dependence Scale-revised (EDS-R, french version) 21 items, 7 subscales, scores from 1-6 for each item and scores above 15 by subscale defining EA.
Personality traits | One single evaluation at a single point in time through study completion, an average of 3 months
  The French version of the Big Five Inventory is a 45-item inventory which measures the five broader domains of personality.

SECONDARY OUTCOMES:
Demographics | One single evaluation at a single point in time through study completion, an average of 3 months
  Age, gender and type of work
Sport Practice (sport) | One single evaluation at a single point in time through study completion, an average of 3 months
  The type of sport practiced
Sport Practice (volume) | One single evaluation at a single point in time through study completion, an average of 3 months
  The volume of training (number of hours weekly)
Sport Practice (number of events) | One single evaluation at a single point in time through study completion, an average of 3 months
  The average number of ultra endurance events per year
Sport Practice (fitness certificate) | One single evaluation at a single point in time through study completion, an average of 3 months
  The type of care practitioner consulted for fitness certificate
Eating habits (dietary supplements) | One single evaluation at a single point in time through study completion, an average of 3 months
  The type of dietary supplement used
Eating habits (SCOFF questionnaire) | One single evaluation at a single point in time through study completion, an average of 3 months
  The two last questions of the SCOFF questionnaire (Fat, Food)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided